CLINICAL TRIAL: NCT02730390
Title: Study on the Efficacy and Safety of Oral Probucol Tablets in Patients With Hyperlipidemia - Post-Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical, Inc., Philippines (Industry)
Responsible Party: Sponsor
Other Study IDs: 009-PPA-1001
Record Dates: First submitted 2016-03-28; First posted 2016-04-06 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Probucol Tablets: Target is 3,000 patients in the Philippines diagnosed with hyperlipidemia (including familial hypercholesterolemia and xanthoma).

SUMMARY:
The primary objective of this post marketing surveillance (PMS) is to determine the safety and efficacy of probucol in lowering the level of serum cholesterol in the blood.

DETAILED DESCRIPTION:
This nationwide post marketing surveillance targets to recruit a total of 3,000 patients with hyperlipidemia. Duration of treatment is 60 days. The usual starting dose for Lorelco is 500 mg administered daily, divided into two (2) doses (250mg BID) and given after meals. The dose may be adjusted according to the patient's age and condition. Lipid serum test will be obtained at Day 0 (Baseline). In subjects requiring antihyperlipidemics that fulfill the inclusion criteria, Lorelco 250 BID will be started. There will be 2 follow-up visits after baseline on Day 30 and Day 60. Both lipid serum tests and ECG will be done on these 2 follow-up visits. During each visit the investigator will assess the subject's vital signs and symptoms and check for any adverse events.

The primary outcome of measure is the percentage reduction or increase in total cholesterol and triglycerides from baseline values at Week 0 to Week 4 and Week 8 using the following scale:

Total Cholesterol Triglycerides

1. Markedly reduced
2. Moderately reduced
3. Slightly reduced
4. Unchanged
5. Increased Reduction of ≥ 15% Reduction of ≥ 10% but < 15% Reduction of ≥ 5% but < 10% Change of < 5% Increase of ≥ 5% Reduction of ≥ 30% Reduction of ≥ 20% but < 30% Reduction of ≥ 10% but < 20% Change of < 10% Increase of ≥ 10% The percentage change on the last week of treatment will be the final evaluation.

The secondary outcome is measured by the changes in symptoms and vital signs. Using the following scale:

1. Markedly Improved
2. Improved
3. Slightly Improved
4. Unchanged
5. Aggravated
6. Unknown (not assessable)

Safety will be measured by the incidence of adverse events to be collected.

Overall efficacy and safety will be evaluated to assess the usefulness of Lorelco using the following scale:

1. Very useful
2. Useful
3. Somewhat useful
4. Not useful
5. Unfavorable
6. Unknown (not assessable)

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with hyperlipidemia including familial hypercholesterolemia and xanthoma.

Exclusion Criteria:

None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 3,000 patients in the Philippines with hyperlipidemia (including familial hypercholesterolemia and xanthoma).
Sampling Method: Non-Probability Sample
Enrollment: 3087 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Efficacy - Improvement in serum lipids. | values will be calculated at Day 30
  Percentage changes in total cholesterol and triglycerides from baseline (Day 0) values will be calculated at Day 30 and Day 60.
Efficacy - Improvement in serum lipids. | values will be calculated at Day 60
  Percentage changes in total cholesterol and triglycerides from

SECONDARY OUTCOMES:
Efficacy - Changes in symptoms and vital signs. | overall 60 days
  Assessed by investigator using following scale:
  1. Markedly Improved
  2. Improved
  3. Slightly Improved
  4. Unchanged
  5. Aggravated
  6. Unknown (not assessable)
Safety - Overall Safety will be evaluated to assess the usefulness of the study drug | overall 60 days
  Check for any adverse event and assess the usefulness

IPD SHARING:
Plan to Share IPD: Undecided